CLINICAL TRIAL: NCT06404294
Title: A Randomized Controlled Study of the External Diaphragm Pacemaker Assisted Extubation in Premature Infants With Invasive Mechanical Ventilation
Brief Title: The External Diaphragm Pacemaker Assisted Extubation in Premature Infants With Invasive Mechanical Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wang Jianhui, Attending neonatologist, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240324
Record Dates: First submitted 2024-04-02; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Invasive Mechanical Ventilation; Extubation
Keywords: External Diaphragm Pacemaker; Invasive Mechanical Ventilation; Extubation; Preterm Infants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be performed by someone who are not involved in this study. Outcomes assessor will review the patients' medical record masked for the type of intervention.The investigators performing the final statistic analyses will also be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Diaphragm Pacemaker treatment group (Experimental): On the basis of conventional treatment, the patients in this group were treated with external diaphragm pacemaker for 2 weeks or until extubation.
  Interventions: Device: External Diaphragm Pacemaker treatment
- No External Diaphragm Pacemaker treatment group (No Intervention): The patients in this group were treated with conventional treatment.

INTERVENTIONS:
Device: External Diaphragm Pacemaker treatment — On the basis of conventional treatment, the patients in this group were treated with external diaphragm pacemaker for 2 weeks or until extubation.The treatment process of external diaphragm pacemaker is as follows: Set parameters: pacing frequency: 5-9 times /min, generally starting from 5 times /min, and adjusted according to the tolerance of the child; Pulse frequency 30 hertz; The stimulation intensity generally starts from 2-3. If the respiratory waveform of the child on the machine is not disturbed, it indicates that the child can tolerate it and the intensity can be appropriately increased. Treatment time: generally starts from 5 minutes, the longest is not more than 20 minutes, the frequency of treatment: 1 time/day in the first week, 2 times/day in the second week.
  Arms: External Diaphragm Pacemaker treatment group

SUMMARY:
With the development of perinatal medicine, more and more newborns with respiratory failure can be treated due to the use of respiratory support technology. However, long-term invasive mechanical ventilation treatment can lead to a series of complications such as ventilator-associated pneumonia, atelectasis and air leakage syndrome, and increase the risk of bronchopulmonary dysplasia and neurodevelopmental lag of premature infants. It also leads to longer hospital stays and higher hospital costs. To shorten the invasive mechanical ventilation time and improve the success rate of withdrawal through various ways is the development direction of neonatal mechanical ventilation therapy.

Respiratory muscle atrophy is common and rapid in children receiving invasive mechanical ventilation, and is an important cause of ventilator dependence and withdrawal failure. The diaphragm of newborns is the main respiratory muscle, of which the diaphragm type 1 endurance fiber accounts for only about 30%, far lower than the proportion of about 55% in adults, so the diaphragm of newborns is more prone to fatigue. Previous animal experiments and clinical studies in children and adults have confirmed that diaphragmatic pacing therapy applied to patients with long-term invasive mechanical ventilation can prevent diaphragmatic atrophy, reverse diaphragmatic injury, significantly improve diaphragmatic thickness, improve diaphragmatic anti-fatigue ability, thereby increasing lung ventilation, relieving dyspnea, and achieving the effect of assisted extubation.

The neonatology Department of the Children's Hospital Affiliated to Chongqing Medical University started neonatal external diaphragm pacemaker treatment in 2022, and has completed 1383 cases so far, initially showing the effectiveness and safety of external diaphragm pacemaker treatment in neonatal population. But so far, there is no systematic evaluation of clinical intervention effect of external diaphragm pacemaker treatment on neonatal respiratory failure patients at home and abroad. Based on this, the project team intends to conduct a prospective randomized controlled study to systematically evaluate the safety of external diaphragm pacemaker in preterm infants requiring invasive mechanical ventilation for ≥7 days at 28 to 35 weeks of gestation, and to evaluate the efficacy of external diaphragm pacemaker in adjuvant extubation.

DETAILED DESCRIPTION:
Neonatal respiratory failure is the central or peripheral respiratory dysfunction caused by various reasons, and is an important clinical critical disease of newborns. With the development of perinatal medicine, more and more newborns with respiratory failure can be treated due to the use of respiratory support technology. However, long-term invasive mechanical ventilation treatment can lead to a series of complications such as ventilator-associated pneumonia, atelectasis and air leakage syndrome, and increase the risk of bronchopulmonary dysplasia and neurodevelopmental lag of premature infants. It also leads to longer hospital stays and higher hospital costs. To shorten the invasive mechanical ventilation time and improve the success rate of withdrawal through various ways is the development direction of neonatal mechanical ventilation therapy.

Respiratory muscle atrophy is common and rapid in children receiving invasive mechanical ventilation, and is an important cause of ventilator dependence and withdrawal failure. The diaphragm of newborns is the main respiratory muscle, of which the diaphragm type 1 endurance fiber accounts for only about 30%, far lower than the proportion of about 55% in adults, so the diaphragm of newborns is more prone to fatigue. Studies have shown that phrenic atrophy usually begins within 18-69 hours of invasive mechanical ventilation and progresses at a rate of 4-7% per day.

Previous animal experiments and clinical studies in children and adults have confirmed that diaphragmatic pacing therapy applied to patients with long-term invasive mechanical ventilation can prevent diaphragmatic atrophy, reverse diaphragmatic injury, significantly improve diaphragmatic thickness, improve diaphragmatic anti-fatigue ability, thereby increasing lung ventilation, relieving dyspnea, and achieving the effect of assisted extubation.

In February 1987, the external diaphragm pacemaker independently developed by Chen et al at Sun Yat-sen University of Medical Science was applied to clinical practice, setting a precedent for external diaphragmatic pacing at home and abroad. The basic principle is to perform low-frequency pulse electrical stimulation of the phrenic nerve through the electrodes on the body surface to make the regular contraction and relaxation of the diaphragm and increase the degree of movement of the diaphragm, so as to improve the ventilation function of the patient. In China, Cai et al observed that external diaphragm pacemaker can increase the degree of immediate diaphragm movement in normal people, and significantly increase the degree of immediate movement in patients with chronic obstructive pulmonary disease and the range of diaphragm movement after continuous treatment for 20-30 days, and significantly improve the symptoms of dyspnea.

The neonatology Department of the Children's Hospital Affiliated to Chongqing Medical University started neonatal external diaphragm pacemaker treatment in 2022, and has completed 1383 cases so far, initially showing the effectiveness and safety of external diaphragm pacemaker treatment in neonatal population. But so far, there is no systematic evaluation of clinical intervention effect of external diaphragm pacemaker treatment on neonatal respiratory failure patients at home and abroad. Based on this, the project team intends to conduct a prospective randomized controlled study to systematically evaluate the safety of external diaphragm pacemaker in preterm infants requiring invasive mechanical ventilation for ≥7 days at 28 to 35 weeks of gestation, and to evaluate the efficacy of external diaphragm pacemaker in adjuvant extubation.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants at 28 to 35 weeks.
2. The premature infant whose invasive mechanical ventilation time ≥7 days.
3. Parents sign an informed consent form.

Exclusion Criteria:

1. The premature infant with congenital airway malformation confirmed by chest CT or bronchofiberscopy.
2. The premature infant with congenital genetic metabolic disease.
3. The premature infant with complex congenital heart disease.
4. The premature infant undergoing surgery.
5. The premature infant with severe brain damage.
6. The premature infant with neuromuscular diseases.
7. The premature infant with congenital skin disease, local skin damage or infection.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasive mechanical ventilation time | through study completion, up to 100 days of life
  Time from invasive mechanical ventilation to extubation

SECONDARY OUTCOMES:
Diaphragm geometry and function | through study completion, up to 100 days of life
  Diaphragm ultrasound
Duration of oxygen use | through study completion, up to 100 days of life
  Duration of oxygen use
Incidence of bronchopulmonary dysplasia | through study completion, up to 100 days of life
  Incidence of bronchopulmonary dysplasia
Mortality | through study completion, up to 100 days of life
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, M.D, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Johnson RW, Ng KWP, Dietz AR, Hartman ME, Baty JD, Hasan N, Zaidman CM, Shoykhet M. Muscle atrophy in mechanically-ventilated critically ill children. PLoS One. 2018 Dec 19;13(12):e0207720. doi: 10.1371/journal.pone.0207720. eCollection 2018. PMID 30566470
- [Result] Dassios T, Vervenioti A, Dimitriou G. Respiratory muscle function in the newborn: a narrative review. Pediatr Res. 2022 Mar;91(4):795-803. doi: 10.1038/s41390-021-01529-z. Epub 2021 Apr 19. PMID 33875805
- [Result] Sieck GC, Fournier M, Blanco CE. Diaphragm muscle fatigue resistance during postnatal development. J Appl Physiol (1985). 1991 Aug;71(2):458-64. doi: 10.1152/jappl.1991.71.2.458. PMID 1834623
- [Result] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Result] Grosu HB, Lee YI, Lee J, Eden E, Eikermann M, Rose KM. Diaphragm muscle thinning in patients who are mechanically ventilated. Chest. 2012 Dec;142(6):1455-1460. doi: 10.1378/chest.11-1638. PMID 23364680
- [Result] Francis CA, Hoffer JA, Reynolds S. Ultrasonographic Evaluation of Diaphragm Thickness During Mechanical Ventilation in Intensive Care Patients. Am J Crit Care. 2016 Jan;25(1):e1-8. doi: 10.4037/ajcc2016563. PMID 26724302
- [Result] Zambon M, Beccaria P, Matsuno J, Gemma M, Frati E, Colombo S, Cabrini L, Landoni G, Zangrillo A. Mechanical Ventilation and Diaphragmatic Atrophy in Critically Ill Patients: An Ultrasound Study. Crit Care Med. 2016 Jul;44(7):1347-52. doi: 10.1097/CCM.0000000000001657. PMID 26992064
- [Result] Breuer T, Hatam N, Grabiger B, Marx G, Behnke BJ, Weis J, Kopp R, Gayan-Ramirez G, Zoremba N, Bruells CS. Kinetics of ventilation-induced changes in diaphragmatic metabolism by bilateral phrenic pacing in a piglet model. Sci Rep. 2016 Oct 19;6:35725. doi: 10.1038/srep35725. PMID 27759115
- [Result] Hsin YF, Chen SH, Yu TJ, Huang CC, Chen YH. Effects of transcutaneous electrical diaphragmatic stimulation on respiratory function in patients with prolonged mechanical ventilation. Ann Thorac Med. 2022 Jan-Mar;17(1):14-20. doi: 10.4103/atm.atm_158_21. Epub 2022 Jan 14. PMID 35198044
- [Result] Sotak M, Roubik K, Henlin T, Tyll T. Phrenic nerve stimulation prevents diaphragm atrophy in patients with respiratory failure on mechanical ventilation. BMC Pulm Med. 2021 Oct 8;21(1):314. doi: 10.1186/s12890-021-01677-2. PMID 34625059